CLINICAL TRIAL: NCT04921319
Title: Optimizing Fluid Management Informed by Ultrasound for Patients With Sepsis
Brief Title: De-resuscitation Informed by Ultrasound for Patients With Sepsis
Acronym: DRI-US
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1694487-1
Record Dates: First submitted 2021-04-07; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-03

CONDITIONS: Sepsis; Septic Shock; Sepsis, Severe; Volume Overload
MeSH Terms: conditions — Sepsis; Shock, Septic; Edema

STUDY DESIGN:
Intervention Model Description: Randomized, unblinded clinical trial of 152 critically ill patients with sepsis admitted to the intensive care unit.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VExUS-Guided Arm (Experimental): Will receive 24 hour fluid balance target based on daily VExUS score.
  Interventions: Diagnostic Test: VExUS score
- Usual Care Control Arm (No Intervention): Treating team will be blinded to results of daily VExUS score and will set 24 hour fluid balance target based on usual care.

INTERVENTIONS:
Diagnostic Test: VExUS score — The care team will be informed of the VExUS immediately after the ultrasound is performed and given a suggested target for the following 24 hours as follows:
  * VExUS 0: "The patient will likely tolerate more fluid if clinically needed."
  * VExUS 1: "The patient has evidence of mild venous congestion. The investigators recommend targeting a net neutral or negative fluid balance with diuresis."
  * VExUS 2-3: "The patient has evidence of moderate to severe venous congestion. The investigators recommend targeting a fluid balance of negative 1-2L with diuresis." If the investigator cannot obtain ultrasound images of sufficient quality to calculate VExUS, the care team will be informed that there is no recommendation for that subject on that day.
  Arms: VExUS-Guided Arm

SUMMARY:
Randomized, unblinded clinical trial of 152 critically ill patients with sepsis admitted to the intensive care unit. The primary determine if using the Venous Excess Ultrasound Score (VExUS) to guide fluid deresuscitation in critically ill patients with sepsis reduces net fluid balance at 5 days as compared to usual care.

DETAILED DESCRIPTION:
Physicians can assess venous congestions with point of care ultrasound of intraabdominal veins using the venous excess in ultrasound score (VExUS), which has been shown to predict the harmful effects of volume overload. We seek to determine if VExUS-guided deresuscitation reduces the fluid balance in critically ill patients with sepsis as compared to usual care. This score compiles findings from the inferior vena cava, hepatic vein Doppler waveform, portal vein Doppler waveform, and intrarenal vein Doppler waveform:

Grade 0: IVC < 2cm, normal pattern in flow patterns of hepatic, portal, and intrarenal veins Grade 1: IVC ≥ 2cm, normal patterns or mild abnormalities in flow patterns of hepatic, portal, and intrarenal veins.

Grade 2: IVC ≥ 2cm, severe venous flow pattern in one among hepatic, portal, and intrarenal veins.

Grade 3: IVC ≥ 2cm, severe venous flow pattern in multiple among hepatic, portal, and intrarenal veins.

After informed consent, subjects will be randomized in a 1:1 ratio to the VExUS-guided intervention arm vs control arm. Subjects in both arms will undergo daily ultrasound, and the investigator will calculate the VExUS immediately after ultrasounds are obtained.

ELIGIBILITY:
Inclusion Criteria:

* 1. Must be suspected by the treating physician to have sepsis as the primary cause of their acute illness as exhibited by 2 or more of the following Systemic Inflammatory Response Syndrome (SIRS) criteria:

  1. Temperature of > 38 C or < 36 C
  2. Heart rate of > 90/min
  3. Respiratory rate of > 20/min or PaCO2 < 32 mm Hg
  4. White blood cell count > 12000/mm3 or < 4000/mm3 or >10% immature bands. 2. Known or suspected infection at the time of screening 3. Admission to the ICU for <24 hours

Since approximately 12% of patients ultimately diagnosed with sepsis do not meet SIRS criteria, SIRS negative patients will be eligible for the study if the treating physician makes a clinical diagnosis of severe sepsis or septic shock.

Exclusion Criteria:

1. Patients with conditions that may interfere with portal Doppler assessments such as cirrhosis or portal thrombosis
2. Patients with severe chronic kidney disease (estimated glomerular filtration rate<15 mL/min per 1.73 m2 calculated using the Modified Diet in Renal Disease formula).
3. Age < 18 years
4. Active atrial fibrillation or atrial flutter
5. Hemodynamic instability due to active hemorrhage
6. Acute cerebral vascular event
7. Acute coronary syndrome (excluding elevated troponin thought to be from demand ischemia)
8. Acute pulmonary edema
9. Status asthmaticus
10. Drug overdose
11. Injury from burn or trauma
12. Status epilepticus
13. Indication for immediate surgery
14. Received CPR within 24 hours of enrollment
15. Pregnancy
16. Incarceration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative Fluid Balance at 5 days post ICU discharge or ICU Discharge | At 5 days post ICU admission or ICU discharge, whichever comes first
  Total fluid balance (ins minus outs)

SECONDARY OUTCOMES:
Incidence of Acute Kidney Injury | At 5 days post ICU admission or ICU discharge, whichever comes first
  acute kidney injury as defined by KDIGO criteria
Incidence of respiratory failure | At 5 days post ICU admission or ICU discharge, whichever comes first
  Incidence of respiratory failure defined by intubation rates, ventilator free days, ventilator days, use of non-invasive positive pressure ventilation, and use of high flow oxygen
Change in SOFA score | At 5 days post ICU admission or ICU discharge, whichever comes first
  Change in Sequential Organ Failure Assessment (SOFA) score during study period, on scale of 0-48, with higher values being a worse outcome
28-day and in-hospital mortality | 28 days and during hospital admission up to 24 weeks
  All-cause mortality.
ICU discharge fluid balance | From ICU admission to ICU discharge or 30 days after ICU admission, whichever comes first
  Cumulative admission fluid balance at time of ICU discharge.
Daily Sonographic B Line Measurement | study enrollment to ICU discharge or 5 days post-enrollment, whichever comes first
  Measured by counting sonographic B lines in 16 lung zones

CONTACTS AND LOCATIONS:
Overall Officials: Keith Corl, MD, Principal Investigator — Rhode Island Hospital / The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beaubien-Souligny W, Rola P, Haycock K, Bouchard J, Lamarche Y, Spiegel R, Denault AY. Quantifying systemic congestion with Point-Of-Care ultrasound: development of the venous excess ultrasound grading system. Ultrasound J. 2020 Apr 9;12(1):16. doi: 10.1186/s13089-020-00163-w. PMID 32270297